CLINICAL TRIAL: NCT05834348
Title: Drug Treatment Patterns and Effects for Metastatic Non-small Cell Lung Cancer Patients In NORway (DELINOR)
Brief Title: A Study to Learn About the Effectiveness of Cancer Medicines in Patients With Metastatic Non-small Cell Lung Cancer in Norway.
Acronym: DELINOR
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7461041; DELINOR (Other: Alias Study Number)
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lorlatinib; Crizotinib; brigatinib; ceritinib; alectinib; atezolizumab; Bevacizumab; Paclitaxel; Carboplatin; Docetaxel; Erlotinib Hydrochloride; Gefitinib; Afatinib; dacomitinib; osimertinib; pembrolizumab; Nivolumab; entrectinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Advanced/metastatic non-small cell lung cancer patients
  Interventions: Drug: lorlatinib; Drug: crizotinib; Drug: brigatinib; Drug: ceritinib; Drug: alectinib; Drug: atezolizumab; Drug: bevacizumab; Drug: paclitaxel; Drug: carboplatin; Drug: docetaxel; Drug: erlotinib; Drug: gefitinib; Drug: afatinib; Drug: dacomitinib; Drug: osimertinib; Drug: pembrolizumab; Drug: nivolumab; Drug: entrectinib

INTERVENTIONS:
Drug: lorlatinib — As provided in real world practice
Drug: crizotinib — As provided in real world practice
Drug: brigatinib — As provided in real world practice
Drug: ceritinib — As provided in real world practice
Drug: alectinib — As provided in real world practice
Drug: atezolizumab — As provided in real world practice
Drug: bevacizumab — As provided in real world practice
Drug: paclitaxel — As provided in real world practice
Drug: carboplatin — As provided in real world practice
Drug: docetaxel — As provided in real world practice
Drug: erlotinib — As provided in real world practice
Drug: gefitinib — As provided in real world practice
Drug: afatinib — As provided in real world practice
Drug: dacomitinib — As provided in real world practice
Drug: osimertinib — As provided in real world practice
Drug: pembrolizumab — As provided in real world practice
Drug: nivolumab — As provided in real world practice
Drug: entrectinib — As provided in real world practice

SUMMARY:
The main purpose of the study is to learn about the effectiveness and treatment sequence of lung cancer medicines. This study is performed outside of clinical trials in Norway in patients with metastatic non-small cell lung cancer. Non-small cell lung cancer is a group of lung cancers named for the kinds of cells found in the cancer and how the cells look under a microscope. Metastasis is when the cancer cells spread to other parts of the body.

This study includes patient's data from the database who:

* Are 18 years of age or older.
* Are confirmed to have metastatic non-small cell lung cancer between 01 January 2009 and 31 December 2022.

The study is based on data collection from 3 national health registries:

* The Cancer Registry of Norway (CRN),
* The Norwegian Patient Registry (NPR),
* The Norwegian Drug Registry (NDR).

Data from these registries will be linked at an individual patient level to create a single, unified dataset. The information collected includes:

Diagnosis, cancer stage at diagnosis, date of diagnosis, birth year, type of medicinal treatment, date of treatment start and end, treating hospital, age, gender, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old with histologically confirmed stage IIIb, IIIc, IVa, or IVb NSCLC at the time of diagnosis
2. Received their first NSCLC diagnosis (stage IIIb, IIIc, IVa, or IVb) between 01 January 2009, and latest available year

Exclusion Criteria:

1. Patients ≥ 18 years old with histologically confirmed stage IIIb, IIIc, IVa, or IVb NSCLC at the time of diagnosis who received radiation therapy with curative intent, defined as a radiation dose larger than 50gy
2. If the data include patients diagnosed after 2021, IIIb patients will be excluded due to changes in the guideline. The updated guidelines for 2022 recommends that patients diagnosed with stage IIIb who have surgery with the intent to cure should not have ''curative'' radiation (i.e.: it is not possible to exclude these from the population from 2022).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are patients with advanced/metastatic non-small cell lung cancer in the Norwegian National cancer registry.
Sampling Method: Non-Probability Sample
Enrollment: 5279 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Norway, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of eligible participants with non-small cell lung cancer (NSCLC) with age greater than (>) 18 years at the time of initiating anticancer therapy was collected retrospectively from the 3 national registries: Cancer Registry of Norway (CRN), the Norwegian Drug Registry (NDR) and the Norwegian Patient Registry (NPR) between 1-Jan-2015, and 31-Dec-2022 (maximum up to 96 months). The study was conducted in Norway.
Pre-assignment Details: Available data was evaluated as per the study objectives, from 23-Jun-2023 to 23-Jan-2024 (approximately 7 months) in this retrospective observational study.
Groups:
- Biomarker Cohort: Participants with NSCLC who were positive for biomarkers (epidermal growth factor [EGFR] or anaplastic lymphoma kinase [ALK] or ROS proto-oncogene 1 [ROS1]) and were identified from CRN, NDR or NPR between 01-Jan-2015 to 31-Dec-2022 were included in this retrospective observational study.
- Non-biomarker Cohort: Participants with NSCLC with unknown biomarker status (EGFR or ALK or ROS1) and were identified from CRN, NDR or NPR between 01-Jan-2015 to 31-Dec-2022 were included in this retrospective observational study.
Period: Overall Study
Arm/Group | Biomarker Cohort | Non-biomarker Cohort
Started | 618 | 4661
Completed | 618 | 4661
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data was retrieved and observed in this retrospective observational study.
Groups:
- Biomarker Cohort: Participants with NSCLC who were positive for biomarkers (EGFR or ALK or ROS1) and were identified from CRN, NDR or NPR between 01-Jan-2015 to 31-Dec-2022 were included in this retrospective observational study.
- Total: Total of all reporting groups
Arm/Group | Biomarker Cohort | Non-biomarker Cohort | Total
Number analyzed (Participants) | 618 | 4661 | 5279
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at diagnosis reported.
  Years | 67.1 (13) | 70.7 (9.7) | 70.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 385 | 2158 | 2543
  Male | 233 | 2503 | 2736
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Duration of Treatment of Anti-cancer Drugs
Description: The duration of treatment of anti-cancer drugs was calculated as median time to treatment (mToT) for first line treatment and the median total ToT for all treatment lines (mTToT) for the anticancer therapies for EGFR+, ALK+ and ROS1+ and was presented in this outcome measure. mToT measured the time on the treatment participants receive as first line treatment, measuring the time from they start the treatment until they stop the first line treatment (or end of follow up), using the Kaplan Meier estimator. mTToT measured the time on all treatment - from the time they start first line treatment, until the point they stop their last treatment line (or end of follow up), using the Kaplan Meier estimator.
Time Frame: From treatment initiation (1-Jan-2015) to end of follow-up (31-Dec-2022) [maximum up to 96 months]; retrospective data was retrieved and analyzed during 7 months of this observational study
Population: Analysis population included all eligible participants whose data was retrieved and observed in this retrospective observational study. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Biomarker Cohort | Non-biomarker Cohort
Number analyzed (Participants) | 398 | 49
Months
  EGFR+ participants receiving osimertinib: mToT: number analyzed (Participants) | 103 | 0
  EGFR+ participants receiving osimertinib: mToT | 11 [10.1 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of participants with events. |
  EGFR+ participants receiving osimertinib: mTToT: number analyzed (Participants) | 103 | 0
  EGFR+ participants receiving osimertinib: mTToT | 14 [11.1 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. |
  EGFR+ participants receiving other TKI: mToT: number analyzed (Participants) | 185 | 0
  EGFR+ participants receiving other TKI: mToT | 9.4 [8.2 to 11.2] |
  EGFR+ participants receiving other TKI: mTToT: number analyzed (Participants) | 185 | 0
  EGFR+ participants receiving other TKI: mTToT | 15.8 [13.7 to 18.1] |
  ALK+ participants receiving alectinib: mToT: number analyzed (Participants) | 55 | 0
  ALK+ participants receiving alectinib: mToT | 20 [14.7 to 23.7] |
  ALK+ participants receiving alectinib: mTToT: number analyzed (Participants) | 55 | 0
  ALK+ participants receiving alectinib: mTToT | 28 [18 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. |
  ALK+ participants receiving brigatinib: mToT: number analyzed (Participants) | 21 | 0
  ALK+ participants receiving brigatinib: mToT | 11 [4.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. |
  ALK+ participants receiving brigatinib: mTToT: number analyzed (Participants) | 21 | 0
  ALK+ participants receiving brigatinib: mTToT | 16 [11.1 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. |
  ALK+ participants receiving crizotinib: mToT: number analyzed (Participants) | 29 | 0
  ALK+ participants receiving crizotinib: mToT | 7 [2.9 to 21.6] |
  ALK+ participants receiving crizotinib: mTToT: number analyzed (Participants) | 29 | 0
  ALK+ participants receiving crizotinib: mTToT | 19 [10.5 to 37.0] |
  ROS1+ participants receiving crizotinib: mToT: number analyzed (Participants) | 5 | 0
  ROS1+ participants receiving crizotinib: mToT | 5 [2.4 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. |
  ROS1+ participants receiving crizotinib: mTToT: number analyzed (Participants) | 5 | 0
  ROS1+ participants receiving crizotinib: mTToT | 18 [4.9 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. |
  Non-biomarker participants receiving crizotinib: mToT: number analyzed (Participants) | 0 | 23
  Non-biomarker participants receiving crizotinib: mToT |  | 3 [2.6 to 13.3]
  Non-biomarker participants receiving crizotinib: mTToT: number analyzed (Participants) | 0 | 23
  Non-biomarker participants receiving crizotinib: mTToT |  | 8.1 [5.6 to 18.8]
  Non-biomarker participants receiving erlotinib: mToT: number analyzed (Participants) | 0 | 26
  Non-biomarker participants receiving erlotinib: mToT |  | 0.9 [0.9 to 6.5]
  Non-biomarker participants receiving erlotinib: mTToT: number analyzed (Participants) | 0 | 26
  Non-biomarker participants receiving erlotinib: mTToT |  | 6.3 [3.7 to 26.7]

2. Primary Outcome: Number of Participants Classified According to Treatments of Anti-cancer Drugs
Description: Number of participants were classified and reported according to the Anti-cancer drugs received during first-line, second-line and third-line treatment after diagnosis of NSCLC.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data was retrieved and observed in this retrospective observational study. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure; "Number Analyzed" signifies participants evaluable for specified rows. All participants under "Number of Participants Analyzed" contributed data to the table but may not have evaluable data for every row.
Measure: Count of Participants; unit: Participants
Arm/Group | Biomarker Cohort | Non-biomarker Cohort
Number analyzed (Participants) | 618 | 2656
Participants
  EGFR+ participants receiving osimertinib in first line: number analyzed (Participants) | 335 | 0
  EGFR+ participants receiving osimertinib in first line | 104 |
  EGFR+ participants receiving gefitinib in first line: number analyzed (Participants) | 335 | 0
  EGFR+ participants receiving gefitinib in first line | 86 |
  EGFR+ participants receiving erlotinib in first line: number analyzed (Participants) | 335 | 0
  EGFR+ participants receiving erlotinib in first line | 50 |
  EGFR+ participants receiving crizotinib in first line: number analyzed (Participants) | 335 | 0
  EGFR+ participants receiving crizotinib in first line | 2 |
  EGFR+ participants receiving other drugs in first line: number analyzed (Participants) | 335 | 0
  EGFR+ participants receiving other drugs in first line | 93 |
  EGFR+ participants receiving IO and/or ChT in second line: number analyzed (Participants) | 139 | 0
  EGFR+ participants receiving IO and/or ChT in second line | 53 |
  EGFR+ participants receiving osimertinib in second line: number analyzed (Participants) | 139 | 0
  EGFR+ participants receiving osimertinib in second line | 25 |
  EGFR+ participants receiving afatinib in second line: number analyzed (Participants) | 139 | 0
  EGFR+ participants receiving afatinib in second line | 22 |
  EGFR+ participants receiving erlotinib in second line: number analyzed (Participants) | 139 | 0
  EGFR+ participants receiving erlotinib in second line | 19 |
  EGFR+ participants receiving other drugs in second line: number analyzed (Participants) | 139 | 0
  EGFR+ participants receiving other drugs in second line | 20 |
  EGFR+ participants receiving IO and/or ChT in third line: number analyzed (Participants) | 44 | 0
  EGFR+ participants receiving IO and/or ChT in third line | 17 |
  EGFR+ participants receiving osimertinib in third line: number analyzed (Participants) | 44 | 0
  EGFR+ participants receiving osimertinib in third line | 13 |
  EGFR+ participants receiving erlotinib in third line: number analyzed (Participants) | 44 | 0
  EGFR+ participants receiving erlotinib in third line | 3 |
  EGFR+ participants receiving other drugs in third line: number analyzed (Participants) | 44 | 0
  EGFR+ participants receiving other drugs in third line | 11 |
  ALK+ participants receiving alecitinib in first line: number analyzed (Participants) | 115 | 0
  ALK+ participants receiving alecitinib in first line | 55 |
  ALK+ participants receiving crizotinib in first line: number analyzed (Participants) | 115 | 0
  ALK+ participants receiving crizotinib in first line | 29 |
  ALK+ participants receiving brigatinib in first line: number analyzed (Participants) | 115 | 0
  ALK+ participants receiving brigatinib in first line | 21 |
  ALK+ participants receiving other drugs in first line: number analyzed (Participants) | 115 | 0
  ALK+ participants receiving other drugs in first line | 10 |
  ALK+ participants receiving alecitinib in second line: number analyzed (Participants) | 51 | 0
  ALK+ participants receiving alecitinib in second line | 14 |
  ALK+ participants receiving lorlatinib in second line: number analyzed (Participants) | 51 | 0
  ALK+ participants receiving lorlatinib in second line | 12 |
  ALK+ participants receiving crizotinib in second line: number analyzed (Participants) | 51 | 0
  ALK+ participants receiving crizotinib in second line | 4 |
  ALK+ participants receiving other drugs in second line: number analyzed (Participants) | 51 | 0
  ALK+ participants receiving other drugs in second line | 21 |
  ALK+ participants receiving lorlatinib in third line: number analyzed (Participants) | 20 | 0
  ALK+ participants receiving lorlatinib in third line | 6 |
  ALK+ participants receiving alectinib in third line: number analyzed (Participants) | 20 | 0
  ALK+ participants receiving alectinib in third line | 4 |
  ALK+ participants receiving crizotinib in third line: number analyzed (Participants) | 20 | 0
  ALK+ participants receiving crizotinib in third line | 2 |
  ALK+ participants receiving other drugs in third line: number analyzed (Participants) | 20 | 0
  ALK+ participants receiving other drugs in third line | 8 |
  ROS1+ participants receiving IO/ChT in first line: number analyzed (Participants) | 22 | 0
  ROS1+ participants receiving IO/ChT in first line | 13 |
  ROS1+ participants receiving crizotinib in first line: number analyzed (Participants) | 22 | 0
  ROS1+ participants receiving crizotinib in first line | 5 |
  ROS1+ participants receiving other drugs in first line: number analyzed (Participants) | 22 | 0
  ROS1+ participants receiving other drugs in first line | 4 |
  ROS1+ participants receiving crizotinib in second line: number analyzed (Participants) | 6 | 0
  ROS1+ participants receiving crizotinib in second line | 2 |
  ROS1+ participants receiving other drugs in second line: number analyzed (Participants) | 6 | 0
  ROS1+ participants receiving other drugs in second line | 4 |
  Non-biomarker participants receiving crizotinib in first line: number analyzed (Participants) | 0 | 2589
  Non-biomarker participants receiving crizotinib in first line |  | 23
  Non-biomarker participants receiving erlotinib in first line: number analyzed (Participants) | 0 | 2589
  Non-biomarker participants receiving erlotinib in first line |  | 26
  Non-biomarker participants receiving IO/ChT in first line: number analyzed (Participants) | 0 | 2589
  Non-biomarker participants receiving IO/ChT in first line |  | 2540
  Non-biomarker participants receiving crizotinib in second line: number analyzed (Participants) | 0 | 58
  Non-biomarker participants receiving crizotinib in second line |  | 7
  Non-biomarker participants receiving erlotinib in second line: number analyzed (Participants) | 0 | 58
  Non-biomarker participants receiving erlotinib in second line |  | 13
  Non-biomarker participants receiving IO/ChT in second line: number analyzed (Participants) | 0 | 58
  Non-biomarker participants receiving IO/ChT in second line |  | 22
  Non-biomarker participants receiving other drugs in second line: number analyzed (Participants) | 0 | 58
  Non-biomarker participants receiving other drugs in second line |  | 16
  Non-biomarker participants receiving erlotinib in third line: number analyzed (Participants) | 0 | 9
  Non-biomarker participants receiving erlotinib in third line |  | 1
  Non-biomarker participants receiving other drugs in third line: number analyzed (Participants) | 0 | 9
  Non-biomarker participants receiving other drugs in third line |  | 8

3. Primary Outcome: Number of Participants Classified According to Treatment Lines of Anti-cancer Drugs
Description: Number of participants were classified and reported according to the treatment lines received including first-line, second-line and third-line treatment after diagnosis of NSCLC.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data was retrieved and observed in this retrospective observational study. Here, "Number Analyzed" signifies number evaluable for specified rows. All participants under "Number of Participants Analyzed" contributed data to the table but may not have evaluable data for every row.
Measure: Count of Participants; unit: Participants
Arm/Group | Biomarker Cohort | Non-biomarker Cohort
Number analyzed (Participants) | 618 | 4661
Participants
  EGFR+: first line treatment: number analyzed (Participants) | 449 | 0
  EGFR+: first line treatment | 335 |
  EGFR+: second line treatment: number analyzed (Participants) | 335 | 0
  EGFR+: second line treatment | 139 |
  EGFR+: third line treatment: number analyzed (Participants) | 139 | 0
  EGFR+: third line treatment | 44 |
  ALK+: first line treatment: number analyzed (Participants) | 131 | 0
  ALK+: first line treatment | 115 |
  ALK+: second line treatment: number analyzed (Participants) | 115 | 0
  ALK+: second line treatment | 51 |
  ALK+: third line treatment: number analyzed (Participants) | 51 | 0
  ALK+: third line treatment | 20 |
  ROS1+: first line treatment: number analyzed (Participants) | 38 | 0
  ROS1+: first line treatment | 22 |
  ROS1+: second line treatment: number analyzed (Participants) | 22 | 0
  ROS1+: second line treatment | 6 |
  Non-biomarker: first line treatment: number analyzed (Participants) | 0 | 4661
  Non-biomarker: first line treatment |  | 2589
  Non-biomarker: second line treatment: number analyzed (Participants) | 0 | 2589
  Non-biomarker: second line treatment |  | 58
  Non-biomarker: third line treatment: number analyzed (Participants) | 0 | 58
  Non-biomarker: third line treatment |  | 9

4. Primary Outcome: Overall Survival (OS)
Description: OS was defined as time from treatment initiation of anticancer therapy to date of death due to any cause. Analysis was performed by Kaplan-Meier method.
Time Frame: From treatment initiation (1-Jan-2015) to date of death (until 31-Dec-2022) [maximum up to 96 months]; retrospective data was retrieved and analyzed during 7 months of this observational study
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Biomarker Cohort | Non-biomarker Cohort
Number analyzed (Participants) | 618 | 4661
Months
  All participants: 2015-2019: number analyzed (Participants) | 298 | 2639
  All participants: 2015-2019 | 19 [16.5 to 21.2] | 5 [4.9 to 5.8]
  All participants: 2020-2022: number analyzed (Participants) | 320 | 2022
  All participants: 2020-2022 | 23 [19.5 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 7 [5.8 to 7.0]
  EGFR+ participants: 2015-2019: number analyzed (Participants) | 229 | 0
  EGFR+ participants: 2015-2019 | 18 [15.3 to 19.3] |
  EGFR+ participants: 2020-2022: number analyzed (Participants) | 220 | 0
  EGFR+ participants: 2020-2022 | 23 [15.6 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. |
  ALK+ participants: 2015-2019: number analyzed (Participants) | 68 | 0
  ALK+ participants: 2015-2019 | 24 [17.4 to 54.7] |
  ALK+ participants: 2020-2022: number analyzed (Participants) | 63 | 0
  ALK+ participants: 2020-2022 | NA [23.3 to NA] — The Median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. |
  ROS+ participants: 2015-2019: number analyzed (Participants) | 38 | 0
  ROS+ participants: 2015-2019 | NA [NA to NA] — The Median, lower and upper limit of 95% CI was not estimable due to insufficient number of participants with events. |
  ROS+ participants: 2020-2022: number analyzed (Participants) | 38 | 0
  ROS+ participants: 2020-2022 | NA [NA to NA] — The Median, lower and upper limit of 95% CI was not estimable due to insufficient number of participants with events. |

5. Secondary Outcome: Percentage of Participants Classified According to the Disease Stage at the Time of Diagnosis
Description: The percentage of participants classified according to the disease stages as 3B, 3C, 4A and 4B at the time of diagnosis were reported in this outcome measure. Cancer stages were classified based on tumor size (T), metastasis to nearby lymph nodes (LN) [N] and distant metastasis (M). Stages were 3B, 3C, 4A and 4B. Stage 3B (T1N3M0, T2N3M0, T3N3M0 and T4N2M0). Stage 3C (T3N3M0, T4N3M0), Stage 4A (anyT, anyM and M1a/M1b), Stage 4B (anyT, anyM and M1c). where T1=<3 cm; T2= 3 to <5 cm; T3= 5 to <7 cm; T4= >7cm. N0=not spread to LN; N1=spread to 1 to 3; N2=spread to 4 to 9; N3=spread >10 axillary LN. M0= no metastasis; M1a= cancer has spread to other lung; M1b= cancer has as a single tumor outside of the chest, such as to a distant lymph node or an organ such as the liver, bones, or brain; M1c= cancer has spread as more than one tumor outside the chest, such as to distant lymph nodes and/or to other organs such as the liver, bones, or brain.
Time Frame: At time of diagnosis (up to 3 months prior to treatment initiation); retrospective data was retrieved and analyzed during 7 months of this observational study
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Biomarker Cohort | Non-biomarker Cohort
Number analyzed (Participants) | 618 | 4661
Percentage of participants
  Stage 3B | 3.5 | 5.6
  Stage 3C | 1.6 | 3.1
  Stage 4A | 36.2 | 36.2
  Stage 4B | 58.6 | 55.1

6. Secondary Outcome: Percentage of Participants Classified According to the NSCLC Histopathological Subtype
Description: Percentage of participants classified according to the NSCLC histopathological subtype viz adenocarcinoma, non-small cell carcinoma, large cell neuroendocrine carcinoma were reported in this outcome measure.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Biomarker Cohort | Non-biomarker Cohort
Number analyzed (Participants) | 618 | 4661
Percentage of participants
  Adenocarcinoma | 94.7 | 80.8
  Non-small cell carcinoma | 5.0 | 16.8
  Large cell neuroendocrine carcinoma | 0.3 | 2.4

7. Secondary Outcome: Number of Participants Classified According to the Selected Participant Administered Non-Cancer Drugs
Description: Number of participants classified according to the selected administered non-cancer drugs (anticoagulants and statins) were reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Biomarker Cohort | Non-biomarker Cohort
Number analyzed (Participants) | 618 | 4661
Participants
  Anticoagulant: Warfarin | 1 | 33
  Anticoagulant: Heparin | 6 | 42
  Anticoagulant: Dalteparin | 99 | 659
  Anticoagulant: Enoxaparin | 79 | 523
  Anticoagulant: Clopidogrel | 12 | 139
  Anticoagulant: Acetylsalicylic acid | 91 | 843
  Anticoagulant: Dipyridamole | 5 | 41
  Anticoagulant: Prasugrel | 1 | 8
  Anticoagulant: Ticagrelor | 2 | 14
  Anticoagulant: Combinations, acetylsalicylic acid | 0 | 48
  Anticoagulant: Dabigatran etexilate | 2 | 28
  Anticoagulant: Rivaroxaban | 14 | 103
  Anticoagulant: Apixaban | 107 | 498
  Anticoagulant: Edoxaban | 15 | 55
  Anticoagulant: Fondaparinux | 0 | 2
  Statin: Simvastatin | 47 | 375
  Statin: Pravastatin | 10 | 34
  Statin: Fluvastatin | 1 | 7
  Statin: Atorvastatin | 97 | 646
  Statin: Rosuvastatin | 11 | 59

8. Secondary Outcome: Number of Packs Dispensed at the Time of Dispensing
Description: Number of packs dispensed to participants at the time of dispensing were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data was retrieved and observed in this retrospective observational study. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable for specified rows. All participants under "Number of Participants Analyzed" contributed data to the table but may not have evaluable data for every row.
Measure: Count of Participants; unit: Participants
Arm/Group | Biomarker Cohort | Non-biomarker Cohort
Number analyzed (Participants) | 618 | 162
Participants
  Alectinib: 1 pack at first dispensation: number analyzed (Participants) | 73 | 0
  Alectinib: 1 pack at first dispensation | 71 |
  Alectinib: 1 pack at second dispensation: number analyzed (Participants) | 69 | 0
  Alectinib: 1 pack at second dispensation | 64 |
  Alectinib: 1 pack at third dispensation: number analyzed (Participants) | 62 | 0
  Alectinib: 1 pack at third dispensation | 51 |
  Alectinib: 1 pack at fourth dispensation: number analyzed (Participants) | 60 | 0
  Alectinib: 1 pack at fourth dispensation | 49 |
  Alectinib: 2 packs at first dispensation: number analyzed (Participants) | 73 | 0
  Alectinib: 2 packs at first dispensation | 1 |
  Alectinib: 2 packs at second dispensation: number analyzed (Participants) | 69 | 0
  Alectinib: 2 packs at second dispensation | 3 |
  Alectinib: 2 packs at third dispensation: number analyzed (Participants) | 62 | 0
  Alectinib: 2 packs at third dispensation | 9 |
  Alectinib: 2 packs at fourth dispensation: number analyzed (Participants) | 60 | 0
  Alectinib: 2 packs at fourth dispensation | 8 |
  Alectinib: 3 packs at first dispensation: number analyzed (Participants) | 73 | 0
  Alectinib: 3 packs at first dispensation | 1 |
  Alectinib: 3 packs at second dispensation: number analyzed (Participants) | 69 | 0
  Alectinib: 3 packs at second dispensation | 2 |
  Alectinib: 3 packs at third dispensation: number analyzed (Participants) | 62 | 0
  Alectinib: 3 packs at third dispensation | 2 |
  Alectinib: 3 packs at fourth dispensation: number analyzed (Participants) | 60 | 0
  Alectinib: 3 packs at fourth dispensation | 3 |
  Alectinib: 4 packs or more at first dispensation: number analyzed (Participants) | 73 | 0
  Alectinib: 4 packs or more at first dispensation | 0 |
  Alectinib: 4 packs or more at second dispensation: number analyzed (Participants) | 69 | 0
  Alectinib: 4 packs or more at second dispensation | 0 |
  Alectinib: 4 packs or more at third dispensation: number analyzed (Participants) | 62 | 0
  Alectinib: 4 packs or more at third dispensation | 0 |
  Alectinib: 4 packs or more at fourth dispensation: number analyzed (Participants) | 60 | 0
  Alectinib: 4 packs or more at fourth dispensation | 0 |
  Osimertinib: 1 pack at first dispensation: number analyzed (Participants) | 142 | 0
  Osimertinib: 1 pack at first dispensation | 131 |
  Osimertinib: 1 pack at second dispensation: number analyzed (Participants) | 126 | 0
  Osimertinib: 1 pack at second dispensation | 102 |
  Osimertinib: 1 pack at third dispensation: number analyzed (Participants) | 114 | 0
  Osimertinib: 1 pack at third dispensation | 86 |
  Osimertinib: 1 pack at fourth dispensation: number analyzed (Participants) | 100 | 0
  Osimertinib: 1 pack at fourth dispensation | 74 |
  Osimertinib: 2 packs at first dispensation: number analyzed (Participants) | 142 | 0
  Osimertinib: 2 packs at first dispensation | 6 |
  Osimertinib: 2 packs at second dispensation: number analyzed (Participants) | 126 | 0
  Osimertinib: 2 packs at second dispensation | 17 |
  Osimertinib: 2 packs at third dispensation: number analyzed (Participants) | 114 | 0
  Osimertinib: 2 packs at third dispensation | 18 |
  Osimertinib: 2 packs at fourth dispensation: number analyzed (Participants) | 100 | 0
  Osimertinib: 2 packs at fourth dispensation | 21 |
  Osimertinib: 3 packs at first dispensation: number analyzed (Participants) | 142 | 0
  Osimertinib: 3 packs at first dispensation | 5 |
  Osimertinib: 3 packs at second dispensation: number analyzed (Participants) | 126 | 0
  Osimertinib: 3 packs at second dispensation | 6 |
  Osimertinib: 3 packs at third dispensation: number analyzed (Participants) | 114 | 0
  Osimertinib: 3 packs at third dispensation | 9 |
  Osimertinib: 3 packs at fourth dispensation: number analyzed (Participants) | 100 | 0
  Osimertinib: 3 packs at fourth dispensation | 4 |
  Osimertinib: 4 packs or more at first dispensation: number analyzed (Participants) | 142 | 0
  Osimertinib: 4 packs or more at first dispensation | 0 |
  Osimertinib: 4 packs or more at second dispensation: number analyzed (Participants) | 126 | 0
  Osimertinib: 4 packs or more at second dispensation | 1 |
  Osimertinib: 4 packs or more at third dispensation: number analyzed (Participants) | 114 | 0
  Osimertinib: 4 packs or more at third dispensation | 1 |
  Osimertinib: 4 packs or more at fourth dispensation: number analyzed (Participants) | 100 | 0
  Osimertinib: 4 packs or more at fourth dispensation | 1 |
  Erlotinib: <1 pack at first dispensation: number analyzed (Participants) | 0 | 40
  Erlotinib: <1 pack at first dispensation |  | 14
  Erlotinib: <1 pack at second dispensation: number analyzed (Participants) | 0 | 21
  Erlotinib: <1 pack at second dispensation |  | 1
  Erlotinib: <1 pack at third dispensation: number analyzed (Participants) | 0 | 11
  Erlotinib: <1 pack at third dispensation |  | 1
  Erlotinib: <1 pack at fourth dispensation: number analyzed (Participants) | 0 | 7
  Erlotinib: <1 pack at fourth dispensation |  | 0
  Erlotinib: 1 pack at first dispensation: number analyzed (Participants) | 72 | 40
  Erlotinib: 1 pack at first dispensation | 65 | 23
  Erlotinib: 1 pack at second dispensation: number analyzed (Participants) | 69 | 21
  Erlotinib: 1 pack at second dispensation | 61 | 15
  Erlotinib: 1 pack at third dispensation: number analyzed (Participants) | 66 | 11
  Erlotinib: 1 pack at third dispensation | 57 | 7
  Erlotinib: 1 pack at fourth dispensation: number analyzed (Participants) | 55 | 7
  Erlotinib: 1 pack at fourth dispensation | 44 | 5
  Erlotinib: 2 packs at first dispensation: number analyzed (Participants) | 72 | 40
  Erlotinib: 2 packs at first dispensation | 4 | 2
  Erlotinib: 2 packs at second dispensation: number analyzed (Participants) | 69 | 21
  Erlotinib: 2 packs at second dispensation | 3 | 3
  Erlotinib: 2 packs at third dispensation: number analyzed (Participants) | 66 | 11
  Erlotinib: 2 packs at third dispensation | 4 | 1
  Erlotinib: 2 packs at fourth dispensation: number analyzed (Participants) | 55 | 7
  Erlotinib: 2 packs at fourth dispensation | 9 | 1
  Erlotinib: 3 packs at first dispensation: number analyzed (Participants) | 72 | 40
  Erlotinib: 3 packs at first dispensation | 3 | 1
  Erlotinib: 3 packs at second dispensation: number analyzed (Participants) | 69 | 21
  Erlotinib: 3 packs at second dispensation | 5 | 2
  Erlotinib: 3 packs at third dispensation: number analyzed (Participants) | 66 | 11
  Erlotinib: 3 packs at third dispensation | 5 | 1
  Erlotinib: 3 packs at fourth dispensation: number analyzed (Participants) | 55 | 7
  Erlotinib: 3 packs at fourth dispensation | 2 | 0
  Erlotinib: 4 packs or more at first dispensation: number analyzed (Participants) | 72 | 40
  Erlotinib: 4 packs or more at first dispensation | 0 | 0
  Erlotinib: 4 packs or more at second dispensation: number analyzed (Participants) | 69 | 21
  Erlotinib: 4 packs or more at second dispensation | 0 | 0
  Erlotinib: 4 packs or more at third dispensation: number analyzed (Participants) | 66 | 11
  Erlotinib: 4 packs or more at third dispensation | 0 | 1
  Erlotinib: 4 packs or more at fourth dispensation: number analyzed (Participants) | 55 | 7
  Erlotinib: 4 packs or more at fourth dispensation | 0 | 1
  Crizotinib: 1 pack at first dispensation: number analyzed (Participants) | 44 | 30
  Crizotinib: 1 pack at first dispensation | 41 | 28
  Crizotinib: 1 pack at second dispensation: number analyzed (Participants) | 36 | 25
  Crizotinib: 1 pack at second dispensation | 31 | 24
  Crizotinib: 1 pack at third dispensation: number analyzed (Participants) | 27 | 17
  Crizotinib: 1 pack at third dispensation | 21 | 15
  Crizotinib: 1 pack at fourth dispensation: number analyzed (Participants) | 26 | 11
  Crizotinib: 1 pack at fourth dispensation | 19 | 10
  Crizotinib: 2 packs at first dispensation: number analyzed (Participants) | 44 | 30
  Crizotinib: 2 packs at first dispensation | 2 | 2
  Crizotinib: 2 packs at second dispensation: number analyzed (Participants) | 36 | 25
  Crizotinib: 2 packs at second dispensation | 4 | 1
  Crizotinib: 2 packs at third dispensation: number analyzed (Participants) | 27 | 17
  Crizotinib: 2 packs at third dispensation | 6 | 2
  Crizotinib: 2 packs at fourth dispensation: number analyzed (Participants) | 26 | 11
  Crizotinib: 2 packs at fourth dispensation | 4 | 1
  Crizotinib: 3 packs at first dispensation: number analyzed (Participants) | 44 | 30
  Crizotinib: 3 packs at first dispensation | 8 | 0
  Crizotinib: 3 packs at second dispensation: number analyzed (Participants) | 36 | 25
  Crizotinib: 3 packs at second dispensation | 7 | 0
  Crizotinib: 3 packs at third dispensation: number analyzed (Participants) | 27 | 17
  Crizotinib: 3 packs at third dispensation | 4 | 0
  Crizotinib: 3 packs at fourth dispensation: number analyzed (Participants) | 26 | 11
  Crizotinib: 3 packs at fourth dispensation | 7 | 0

9. Secondary Outcome: Number of Participants Classified as Per Specific Norwegian Health Regions
Description: Number of participants classified according to the Norwegian health regions were reported in this outcome measure.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Biomarker Cohort | Non-biomarker Cohort
Number analyzed (Participants) | 618 | 4661
Participants
  Central Norway Regional Health Authority | 70 | 665
  Northern Norway Regional Health Authority | 44 | 488
  South-East Norway Regional Health Authority | 341 | 2427
  Western Norway Regional Health Authority | 156 | 1055
  Unknown | 7 | 26

ADVERSE EVENTS:
Time Frame: All-cause mortality: From treatment initiation (1-Jan-2015) to end of follow-up (31-Dec-2022) [maximum up to 96 months]; retrospective data was retrieved and analyzed during 7 months of this observational study. For adverse events it was not applicable as adverse event data was not planned to be assessed
Description: This study is retrospective, it involves data that exist as structured data by the time of study start. From data source, individual participant data were not retrieved or validated. The minimum criteria for reporting an adverse event (AE) (i.e., identifiable participant, identifiable reporter, a suspect product, and event) cannot be met. Hence, adverse events were not planned to be assessed and are not reported.
Arm/Group | Biomarker Cohort | Non-biomarker Cohort
All-Cause Mortality (participants affected / at risk) | 364/618 | 3780/4661
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The observation period was changed from 1-Jan-2009 to 1-Jan-2015 based on sponsor decision as only a few participants with uncertain about the data quality were recorded prior 2015.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT05834348/Prot_SAP_000.pdf